CLINICAL TRIAL: NCT02207621
Title: A Double-masked, Randomized, Multi-center, Active-controlled, Parallel, 12-month Study Assessing the Safety and Ocular Hypotensive Efficacy of AR-13324 Ophthalmic Solution, 0.02% q.d. and b.i.d. Compared to Timolol Maleate Ophthalmic Solution, 0.5% b.i.d. in Patients With Elevated Intraocular Pressure
Brief Title: Evaluation of Netarsudil (AR-13324) Ophthalmic Solution in Patients With Glaucoma and Ocular Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Aerie Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AR-13324-CS302
Record Dates: First submitted 2014-07-31; First posted 2014-08-04 (Estimated); Results first posted 2018-04-06 (Actual); Last update posted 2018-04-06 (Actual); Status verified 2018-01

CONDITIONS: Ocular Hypertension; Open-angle Glaucoma
Keywords: Glaucoma
MeSH Terms: conditions — Ocular Hypertension; Glaucoma, Open-Angle; Glaucoma | interventions — netarsudil; BID protein, human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- AR-13324 Ophthalmic Solution 0.02% & placebo (Experimental): 1 drop AR-13324 in the evening (PM) & 1 drop placebo in the morning (AM) in both eyes (OU)
  Interventions: Drug: AR-13324 Ophthalmic Solution 0.02%; Other: Placebo
- Timolol maleate Ophthalmic Solution 0.5% BID (Active Comparator): 1 drop twice daily (BID) in the morning (AM) and evening (PM) in both eyes (OU)
  Interventions: Drug: Timolol maleate Ophthalmic Solution 0.5% BID
- AR-13324 Ophthalmic Solution 0.02% BID (Experimental): 1 drop AR-13324 twice daily (BID) in the morning (AM) and evening (PM) in both eyes (OU)
  Interventions: Drug: AR-13324 Ophthalmic Solution 0.02% BID

INTERVENTIONS:
Drug: AR-13324 Ophthalmic Solution 0.02% — 1 drop once daily (QD), PM, OU
  Other Names: Netarsudil
  Arms: AR-13324 Ophthalmic Solution 0.02% & placebo
Drug: Timolol maleate Ophthalmic Solution 0.5% BID — 1 drop BID, AM/PM, OU
  Arms: Timolol maleate Ophthalmic Solution 0.5% BID
Other: Placebo — 1 drop QD, AM, OU
  Arms: AR-13324 Ophthalmic Solution 0.02% & placebo
Drug: AR-13324 Ophthalmic Solution 0.02% BID — 1 drop BID, AM/PM, OU
  Other Names: Netarsudil
  Arms: AR-13324 Ophthalmic Solution 0.02% BID

SUMMARY:
Evaluation of the ocular hypotensive efficacy and safety of Netarsudil (AR-13324) Ophthalmic Solution compared to Timolol Maleate Ophthalmic Solution

ELIGIBILITY:
Subject inclusion criteria

1. 0-2 years of age and 18 years or greater
2. Diagnosis of open angle glaucoma or ocular hypertension
3. Unmedicated (post-washout) intraocular pressure (IOP) >20 mm Hg and < 27 mm Hg in the study eye at 2 qualification visits
4. Corrected visual acuity in each eye equivalent to 20/200
5. Able and willing to give signed informed consent (parent or guardian consent for pediatric patient) and follow study instructions

Subject exclusion criteria

Ophthalmic:

1. Glaucoma: pseudoexfoliation or pigment dispersion component, history of angle closure, or narrow angles. Note: Previous laser peripheral iridotomy is NOT acceptable.
2. Intraocular pressure ≥27 mm Hg (unmedicated) in both eyes or use of more than two ocular hypotensive medications within 30 days of screening. Note: fixed dose combinations count as two medications.
3. Known hypersensitivity to any component of the formulations to be used (benzalkonium chloride, etc.), to topical anesthetics or beta-adrenoceptor antagonists.
4. Previous glaucoma intraocular surgery or glaucoma laser procedures in either eye
5. Refractive surgery in either eye.
6. Ocular trauma in either eye within the six months prior to screening, or ocular surgery or non-refractive laser treatment within the three months prior to screening.
7. Recent or current evidence of ocular infection or inflammation in either eye. Current evidence of clinically significant blepharitis, conjunctivitis, or a history of herpes simplex or zoster keratitis at screening in either eye.
8. Ocular medication in either eye of any kind within 30 days of screening.
9. Clinically significant ocular disease in either eye (e.g., corneal edema, uveitis, severe keratoconjunctivitis sicca) which might interfere with the study, including glaucomatous damage so severe that washout of ocular hypotensive medications for one month is not judged safe.
10. Central corneal thickness in either eye greater than 600 µm at screening.
11. Any abnormality in either eye preventing reliable applanation tonometry of either eye.

    Systemic:
12. Clinically relevant abnormalities (as determined by the investigator) in laboratory tests at screening which may impact the study.
13. Known hypersensitivity or contraindication to beta-adrenoceptor antagonists (e.g., chronic obstructive pulmonary disease or bronchial asthma; abnormally low blood pressure or heart rate; second or third degree heart block or congestive heart failure; severe diabetes).
14. Clinically significant systemic disease (e.g., uncontrolled diabetes, myasthenia gravis, hepatic, renal, endocrine or cardiovascular disorders) which might interfere with the study.
15. Participation in any investigational study within 30 days prior to screening.
16. Changes of systemic medication that could have an effect on intraocular pressure within 30 days prior to screening, or anticipated during the study.
17. Women of childbearing potential who are pregnant, nursing, planning a pregnancy, or not using a medically acceptable form of birth control. An adult woman is considered to be of childbearing potential unless she is one year post-menopausal or three months post-surgical sterilization. All females of childbearing potential must have a negative urine pregnancy test result at the screening examination and must not intend to become pregnant during the study..

Max Age: 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 756 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Theresa Heah, MD, Study Director — Aerie Pharmaceuticals, Inc.
Locations (1):
- Aerie Pharmaceuticals, Bedminster, New Jersey, United States

REFERENCES:
- [Derived] Mundorf T, Mah F, Sheng H, Heah T. Effects of Netarsudil on the Corneal Endothelium: Three-Month Findings from a Phase 3 Trial. Ophthalmol Glaucoma. 2020 Nov-Dec;3(6):421-425. doi: 10.1016/j.ogla.2020.04.014. Epub 2020 Apr 29. PMID 33250082

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 62 clinical trial sites participated in this study, of which 60 clinical trial sites enrolled participants. Screening started in June 2014. Enrollment started in July 2014. The last participant was enrolled in March 2015.
Pre-assignment Details: Prior to enrollment, adult participants were required to have a Screening Visit and 2 Qualification Visits to allow for washout of ocular hypotensive medication.
Groups:
- AR-13324 Ophthalmic Solution 0.02% & Placebo: 1 drop AR-13324 in the evening (PM) and 1 drop placebo in the morning (AM) in both eyes (OU)
- Timolol Maleate Ophthalmic Solution 0.5% BID: 1 drop Timolol maleate twice daily (BID) in the morning (AM) and evening (PM) in both eyes (OU)
Period: Overall Study
Arm/Group | AR-13324 Ophthalmic Solution 0.02% & Placebo | Timolol Maleate Ophthalmic Solution 0.5% BID | AR-13324 Ophthalmic Solution 0.02% BID
Started | 251 | 251 | 254
Completed | 146 | 204 | 86
Not Completed | 105 | 47 | 168
Not completed — Adverse Event | 71 | 15 | 132
Not completed — Withdrawal by Subject | 9 | 9 | 13
Not completed — Non-Compliant | 3 | 3 | 1
Not completed — Lost to Follow-up | 1 | 0 | 3
Not completed — Lack of Efficacy | 10 | 2 | 4
Not completed — Disallowed Concurrent Medication | 2 | 5 | 2
Not completed — Physician Decision | 1 | 2 | 2
Not completed — Protocol Violation | 4 | 10 | 6
Not completed — Death | 2 | 0 | 0
Not completed — Other(Site,Sponsor and Subject request) | 2 | 1 | 5

BASELINE CHARACTERISTICS:
Population: The randomized population includes all subjects who were randomized to treatment. Baseline variables and demographic characteristics were summarized for this population.
Groups:
- Total: Total of all reporting groups
Arm/Group | AR-13324 Ophthalmic Solution 0.02% & Placebo | Timolol Maleate Ophthalmic Solution 0.5% BID | AR-13324 Ophthalmic Solution 0.02% BID | Total
Number analyzed (Participants) | 251 | 251 | 254 | 756
Age, Continuous [Mean (Standard Deviation); unit: Years] | 65.3 (11.48) | 63 (11.81) | 64.1 (12.46) | 64.1 (11.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 148 | 150 | 165 | 463
  Male | 103 | 101 | 89 | 293
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 41 | 42 | 43 | 126
  Not Hispanic or Latino | 210 | 209 | 211 | 630
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 0 | 2
  Asian | 2 | 6 | 6 | 14
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 69 | 76 | 69 | 214
  White | 178 | 166 | 177 | 521
  More than one race | 0 | 2 | 1 | 3
  Unknown or Not Reported | 0 | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Intraocular Pressure (IOP)
Description: The primary efficacy outcome is mean intraocular pressure (IOP)
Time Frame: 3 months
Population: The Per Protocol (PP) population includes all subjects who did not have a major protocol violation likely to seriously affect the primary outcome of the study. This is the primary population for efficacy analyses.
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- AR-13324 Ophthalmic Solution 0.02% & Placebo: 1 drop AR-13324 in the PM & 1 drop placebo in the AM, OU
- Timolol Maleate Ophthalmic Solution 0.5% BID: 1 drop Timolol maleate BID in the AM and PM, OU
- AR-13324 Ophthalmic Solution 0.02% BID: 1 drop AR-13324 BID in the AM and PM, OU
Arm/Group | AR-13324 Ophthalmic Solution 0.02% & Placebo | Timolol Maleate Ophthalmic Solution 0.5% BID | AR-13324 Ophthalmic Solution 0.02% BID
Number analyzed (Participants) | 206 | 217 | 209
mmHg
  Day 1, 0800 hours | 23.51 (1.654) | 23.45 (1.601) | 23.50 (1.671)
  Day 1, 1000 hours | 22.31 (2.131) | 22.18 (2.089) | 22.26 (2.103)
  Day 1, 1600 hours | 21.56 (2.338) | 21.61 (2.369) | 21.49 (2.279)
  Day 15, 0800 hours | 19.01 (2.979) | 18.25 (2.736) | 18.20 (3.491)
  Day 15, 1000 hours | 17.74 (3.089) | 17.49 (2.796) | 16.91 (3.087)
  Day 15, 1600 hours | 17.37 (2.830) | 17.59 (2.935) | 16.28 (2.925)
  Day 43, 0800 hours | 19.37 (3.749) | 18.08 (2.614) | 18.57 (3.206)
  Day 43, 1000 hours | 18.10 (3.335) | 17.31 (2.805) | 17.09 (3.028)
  Day 43, 1600 hours | 17.88 (2.888) | 17.25 (2.813) | 16.58 (3.095)
  Day 90 (Month 3), 0800 hours | 19.43 (3.761) | 18.21 (2.819) | 18.66 (3.460)
  Day 90 (Month 3), 1000 hours | 18.18 (3.571) | 17.52 (2.777) | 17.81 (3.330)
  Day 90 (Month 3), 1600 hours | 17.73 (3.386) | 17.67 (2.879) | 17.08 (3.112)

2. Secondary Outcome: Extent of Exposure
Description: Exposure to study medication in days for all treatment groups
Time Frame: 12 Months
Population: The Safety Population included all randomized subjects who received at least 1 dose of study medication and was used to summarize safety variables. The safety population summarized subjects as treated for purpose of analysis. One (1) subject did not receive study drug as randomized, shown in the Participant Flow
Measure: Mean (Standard Deviation); unit: days
Groups:
- AR-13324 Ophthalmic Solution 0.02% & Placebo: 1 drop AR-13324 in the PM and 1 drop placebo in the AM in both eyes
Arm/Group | AR-13324 Ophthalmic Solution 0.02% & Placebo | Timolol Maleate Ophthalmic Solution 0.5% BID | AR-13324 Ophthalmic Solution 0.02% BID
Number analyzed (Participants) | 251 | 251 | 253
days | 259.7 (133.34) | 324.5 (90.73) | 185.2 (144.56)

ADVERSE EVENTS:
Time Frame: 1 year
Description: The Safety Population included all randomized subjects who received at least 1 dose of study medication and was used to summarize safety variables. One (1) subject did not receive study drug as randomized, shown in the Participant Flow.
Groups:
- AR-13324 Ophthalmic Solution 0.02% & Placebo: 1 drop AR-13324 in the PM and 1 drop placebo in the AM, OU
Arm/Group | AR-13324 Ophthalmic Solution 0.02% & Placebo | Timolol Maleate Ophthalmic Solution 0.5% BID | AR-13324 Ophthalmic Solution 0.02% BID
All-Cause Mortality (participants affected / at risk) | 2/251 | 0/251 | 0/253
Serious Adverse Events (participants affected / at risk) | 17/251 | 12/251 | 7/253
Other Adverse Events (participants affected / at risk) | 198/251 | 96/251 | 213/253
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AR-13324 Ophthalmic Solution 0.02% & Placebo (N=251) | Timolol Maleate Ophthalmic Solution 0.5% BID (N=251) | AR-13324 Ophthalmic Solution 0.02% BID (N=253)
Coronary Artery Disease (Cardiac disorders) | 2 | 0 | 1
Myocardial Infarction (Cardiac disorders) | 2 | 1 | 1
Atrial Fibrillation (Cardiac disorders) | 2 | 0 | 0
Atrial Flutter (Cardiac disorders) | 1 | 0 | 0
Bradycardia (Cardiac disorders) | 1 | 0 | 0
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Malignant Melanoma in Situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Myelodysplastic Syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Foot Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Postoperative Ileus (Injury, poisoning and procedural complications) | 1 | 0 | 0
Road Traffic Accident (Injury, poisoning and procedural complications) | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0
Hip Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Ligament Rupture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Tendon Rupture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Synovial Cyst (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Cerebrovascular Accident (Nervous system disorders) | 1 | 0 | 0
Embolic Stroke (Nervous system disorders) | 1 | 0 | 0
Carotid Artery Stenosis (Nervous system disorders) | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pulmonary Artery Stenosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Accelerated Hypertension (Vascular disorders) | 1 | 0 | 0
Internal Haemorrhage (Vascular disorders) | 0 | 0 | 1
Peripheral Artery Occlusion (Vascular disorders) | 0 | 1 | 0
Abdominal Pain (Gastrointestinal disorders) | 0 | 0 | 1
Gastric Ulcer Perforation (Gastrointestinal disorders) | 0 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0
Peritonitis Bacterial (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0
Urinary Tract Infection (Infections and infestations) | 0 | 1 | 0
Fluid Overload (Metabolism and nutrition disorders) | 1 | 0 | 0
Acute Kidney Injury (Renal and urinary disorders) | 0 | 1 | 1
Renal Failure (Renal and urinary disorders) | 0 | 1 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Cataract (Eye disorders) | 0 | 1 | 0
Prostatic Specific Antigen Increased (Investigations) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AR-13324 Ophthalmic Solution 0.02% & Placebo (N=251) | Timolol Maleate Ophthalmic Solution 0.5% BID (N=251) | AR-13324 Ophthalmic Solution 0.02% BID (N=253)
Conjunctival Hyperaemia (Eye disorders) | 152 | 35 | 168
Cornea Verticillata (Eye disorders) | 64 | 2 | 64
Conjunctival Haemorrhage (Eye disorders) | 49 | 2 | 49
Vision Blurred (Eye disorders) | 27 | 7 | 44
Lacrimation Increased (Eye disorders) | 19 | 0 | 25
Visual Acuity Reduced (Eye disorders) | 22 | 6 | 22
Eye Pruritus (Eye disorders) | 14 | 3 | 20
Conjunctival Oedema (Eye disorders) | 8 | 0 | 19
Erythema of Eyelid (Eye disorders) | 14 | 2 | 12
Eye Irritation (Eye disorders) | 11 | 8 | 13
Foreign Body Sensation in Eyes (Eye disorders) | 7 | 1 | 14
Instillation Site Pain (General disorders) | 45 | 41 | 45
Instillation Site Erythema (General disorders) | 14 | 5 | 32
Vital Dye Staining Cornea Present (Investigations) | 14 | 14 | 17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No